CLINICAL TRIAL: NCT03680807
Title: Power Production in Older Adults With Knee Osteoarthritis Compared to Healthy Counterparts
Brief Title: Power Production in Older Adults With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Evelien Van Roie, Dr., KU Leuven
Other Study IDs: S60595
Record Dates: First submitted 2018-09-18; First posted 2018-09-21 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Osteo Arthritis Knee
Keywords: Knee osteoarthritis; power production; functional capacity
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Older adults with knee osteoarthritis (>50 years)
  Interventions: Diagnostic Test: Muscle function test
- Healthy older adults (> 50 years)
  Interventions: Diagnostic Test: Muscle function test

INTERVENTIONS:
Diagnostic Test: Muscle function test — Power and strength tests of the knee-extensor muscles, handgrip strength, functional capacity tests

SUMMARY:
Knee osteoarthritis is an important cause of functional disabilities at old age. Previous research has demonstrated that individuals with knee osteoarthritis have reduced knee-extensor strength in comparison to healthy individuals. However, rapid power production declines more than strength as a consequence of ageing and is more predictive of functional capacity. However, limited research has investigated whether individuals with knee osteoarthritis have reduced ability to develop strength and power rapidly on top of reduced maximal strength capacities, which is the primary aim of the current study.

ELIGIBILITY:
Inclusion Criteria:

Group with knee osteoarthritis:

- Diagnosed with knee osteoarthritis based on RX.

Exclusion Criteria:

Healthy group:

* Systematic engagement in (resistance) exercise in the 12-months prior to participation
* Cardiovascular disease
* Neurological disorders
* Cognitive malfunctioning
* Severe knee or hip problems

Group with knee osteoarthritis:

* Systematic engagement in (resistance) exercise in the 12-months prior to participation
* Cardiovascular disease
* Neurological disorders
* Cognitive malfunctioning
* Severe hip problems

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults between 50 and 80 years with or without knee osteoarthritis. Subjects are sedentary or recreationally active.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Rate of power development | up to 3 months
  Subjects perform a test protocol on a Biodex dynamometer, consisting of isotonic contractions of the leg-extensor muscles. Subjects are instructed to kick as fast as possible against different (relative) loads. The rate of power development (watt/s) is defined as the linear slope of the power-time curve and is measured from the onset of movement till peak power.

SECONDARY OUTCOMES:
Maximal isometric strength | up to 3 months
  Maximal strength (Nm) is measured by means of unilateral isometric knee-extensor tests on a Biodex dynamometer.
Maximal isokinetic strength | up to 3 months
  Maximal strength (Nm) is measured by means of unilateral isokinetic knee-extensor tests on a Biodex dynamometer.
Stair Climbing performance | up to 3 months
  Stair ascent duration (in s), the time needed to ascent a flight of stairs.
Gait speed | up to 3 months
  The average speed to walk 10m as fast as possible (in m/s).
5 repetition sit-to-stand test | up to 3 months
  The time needed to perform 5 sit-to-stand transitions (in s).
Timed-up-and-go | up to 3 months
  The time needed to stand up from a chair, walk 3m, turn, walk back and sit down.
Handgrip strength | up to 3 months
  Handgrip strength (kg) evaluated with Jamar dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Movement Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No